CLINICAL TRIAL: NCT05807789
Title: Molecular-genetic Characterization in Patients Undergoing CAR-T Cell Infusion
Acronym: CAR_22
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Francesca Bonifazi, MD, MD, Director of Hematopoietic Stem Cell Transplant Program, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: CAR_22
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hematologic Malignancy
Keywords: CAR-T
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In recent years, the application of increasingly advanced methods of ex-vivo cell culture and cell engineering has made it possible to develop new cellular therapeutic platforms including the "CAR (Chimeric Antigen Receptor) - T cell therapy". CAR-T cell therapy is a therapy that uses T lymphocytes engineered to express a chimeric receptor directed against a specific antigen, theoretically applicable to the treatment of all neoplasms but currently more widely used in the treatment of haematological malignancies. One of the most innovative aspects introduced with CAR-T cell therapy is that of living-drug, cells that act as a drug as well as a means to build specific immunity against the neoplasm. The advantages of this therapy are therefore represented by the possibility of refueling the patient's immunity, deficient in the control of the neoplastic disease, with lymphocytes capable of expressing an antineoplastic activity with mechanisms not subject to restriction of HLA-mediated antigen recognition.

However, the use of CAR-T therapies is not free from potentially serious and sometimes lethal adverse events; in the toxicity profile the following are recognizable as peculiar:

* cytokine release syndrome (CRS)
* B-cell aplasia (hypogammaglobulinemia)
* neurological adverse reactions
* haematological toxicity
* infections. Therefore, considering that on the one hand adverse events are not negligible and on the other hand that a percentage > 50% of patients lose the response obtained, it is necessary to improve the therapeutic profile of CAR-T cell therapy by increasing its efficacy and reducing its toxicity . Both of these strategies are linked to the understanding of the resistance mechanisms of neoplastic cells, as well as to the biology of CAR-T cells and of all the cellular (microenvironment) and non-cellular systems with which they interact.

DETAILED DESCRIPTION:
In recent years, the application of increasingly advanced methods of ex-vivo cell culture and cell engineering has made it possible to develop new cellular therapeutic platforms including the "CAR (Chimeric Antigen Receptor) - T cell therapy". CAR-T cell therapy is a therapy that uses T lymphocytes engineered to express a chimeric receptor directed against a specific antigen, theoretically applicable to the treatment of all neoplasms but currently more widely used in the treatment of haematological malignancies. One of the most innovative aspects introduced with CAR-T cell therapy is that of living-drug, cells that act as a drug as well as a means to build specific immunity against the neoplasm.

The CAR-T cell therapy program is divided into three fundamental points:

* the collection of lymphocytes (by apheresis) destined for the engineering process;
* the manufacturing aimed at transducing and expanding the collected lymphocytes;
* the infusion of cell product after lymphodepleting chemotherapy.

The advantages of this therapy are therefore represented by the possibility of refueling the patient's immunity, deficient in the control of the neoplastic disease, with lymphocytes capable of expressing an antineoplastic activity with mechanisms not subject to restriction of HLA-mediated antigen recognition.

Currently the Marketing Authorization (MA) in the European Union and Italy provides for the use of therapies with anti-CD19 CAR-T cells based on second generation chimeric constructs:

* tisagenlecleucel (Kymriah): pediatric patients and young adults up to 25 years of age included with B-cell acute lymphoblastic leukemia (ALL) that is refractory, relapsing post-transplant or in second or further recurrence; adult patients with diffuse lymphoma a relapsed or refractory large B-cell (DLBCL) after two or more lines of therapy systemic; adult patients with relapsed or refractory follicular lymphoma (LF) after two or more lines of systemic therapy.
* axicabtagene ciloleucel (Yescarta): adult patients with diffuse large lymphoma B-cells (DLBCL) and primary lymphoma of the mediastinum a refractory or relapsing large B-cell (PMBCL) cells, after two or more lines of systemic therapy; adult patients with refractory or relapsed follicular lymphoma (FL) after three or more lines of systemic therapy.
* brexucabtagene autoleucel (Tecartus): adult patients with cell lymphoma mantle disease (MCL) relapsed or refractory after two or more lines of systemic therapy including a Bruton's tyrosine kinase inhibitor. The marketing authorization for lisocabtagene maraleucel (Breyanzi) is expected shortly for the treatment of diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL) and follicular lymphoma (LF) grade 3B, refractory or relapsing.

However, the use of CAR-T therapies is not free from potentially serious and sometimes lethal adverse events; in the toxicity profile the following are recognizable as peculiar:

* cytokine release syndrome (CRS)
* B-cell aplasia (hypogammaglobulinemia)
* neurological adverse reactions
* haematological toxicity
* infections. Therefore, considering that on the one hand adverse events are not negligible and on the other hand that a percentage > 50% of patients lose the response obtained, it is necessary to improve the therapeutic profile of CAR-T cell therapy by increasing its efficacy and reducing its toxicity . Both of these strategies are linked to the understanding of the resistance mechanisms of neoplastic cells, as well as to the biology of CAR-T cells and of all the cellular (microenvironment) and non-cellular systems with which they interact.

The importance of the study lies in the investigations aimed at understanding the possible strategies that allow the neoplastic cell to evade the mechanisms of CAR-T mediated cytotoxicity and/or alter the structure of the antigen, making it functionally "invisible" to the interaction with the CAR ; it will thus be possible to identify mechanisms of resistance to treatment with CAR-T cells. Another strong point of the study is represented by the single cell sequencing to identify subpopulations of lymphoid (CAR+ and CAR-) and myeloid cells related to the clinical outcome (toxicity and response to treatment).

Therefore, the primary objectives of the study are:

* Genomic studies in peripheral blood samples taken from patients affected by hematological malignancies undergoing CAR-T cell therapy, in order to identify correlations between neoplastic cell signatures and response to therapy (evaluated according to laboratory and instrumental standards).
* Study of CAR+ and CAR- lymphoid populations and of myeloid populations with single-cell RNA sequencing platforms in peripheral blood samples in order to understand the cellular dynamics related to clinical outcomes such as response to therapy (evaluated according to laboratory and instrumental standards) and adverse events (CRS, ICANS, sHLH, coagulopathy, cytopenias, and autoimmune dyscrasias).

Tumor profiling will result in the kinetics of the allele frequency of variants specific genes (VAFs) (identified by NGS sequencing of free DNA circulating) in patients with different clinical outcome (response or refractoriness to treatment with CAR-T therapy). Single cell RNA sequencing (scRNAseq) will output gene abundance values and cell clusters (subpopulations of CAR+ and CAR- lymphoid cells and myeloid cells) concomitantly of events considered relevant in the patient's clinical history, such as the occurrence of toxicity and loss or maintenance of response to treatment, in order to establish the possible correlations.

The study will be proposed to all patients aged ≥ 18 years undergoing CAR-T cell infusion at the Departmental Program of Advanced Cellular Therapies of the IRCCS AOU of Bologna, about 50 patients a year for a total of 150 patients.

Peripheral blood samples will be used to perform the study will be picked up at the following times:

* to apheresis;
* on entering the ward;
* per day -1;
* on day 0 (2 h post-infusion);
* per day +1, +3, +5, +7, +9, +11, +13, +30, +90, +180, +365;

The sampling of tissues coincides with the sampling that represent the current standard in routine clinical practice in the patient undergoing CAR-T therapy:

the samples will be obtained without invalidating the assistance procedures (diagnostic-therapeutic) regularly scheduled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years.
2. Patients with haematological pathology hospitalized for CAR-T cell infusion therapeutic program (with Marketing Authorization) at the Departmental Program of Advanced Cellular Therapies, of the IRCCS AOU of Bologna
3. Patients with express consent to participate in this study, acquired by signing the informed consent.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be proposed to all patients aged ≥ 18 years undergoing CAR-T cell infusion at the Departmental Program of Advanced Cellular Therapies of the IRCCS AOU of Bologna
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Genomic studies | 3 years
  Genomic studies in peripheral blood samples taken from patients affected by hematological malignancies undergoing CAR-T cell therapy, in order to identify correlations between neoplastic cell signatures and response to therapy (evaluated according to laboratory and instrumental standards).
Study of CAR+ and CAR- lymphoid populations and of myeloid populations | 3 years
  Study of CAR+ and CAR- lymphoid populations and of myeloid populations with single-cell RNA sequencing platforms in peripheral blood samples in order to understand the cellular dynamics related to clinical outcomes such as response to therapy (evaluated according to laboratory and instrumental standards) and adverse events (CRS, ICANS, sHLH, coagulopathy, cytopenias, and autoimmune dyscrasias).

CONTACTS AND LOCATIONS:
Locations (1):
- Programma Dipartimentale Terapie Cellulari Avanzate, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes